CLINICAL TRIAL: NCT01860326
Title: An Open-label Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Single Oral Doses of DEB025 in Subjects With Mild and Moderate Hepatic Impairment Compared to Matched Healthy Subjects With Normal Liver Function
Brief Title: Evaluate the Pharmacokinetics, Safety, and Tolerability of Alisporivir in Subjects With Hepatic Impairment Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CDEB025A2114
Record Dates: First submitted 2012-02-21; First posted 2013-05-22 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Hepatic Insufficiency
Keywords: hepatic impairment; mild and moderate hepatic impairment; Alisporivir
MeSH Terms: conditions — Hepatic Insufficiency; Lymphoma, Follicular | interventions — alisporivir

ARMS (1):
- Alisporivir (Experimental): Single 200 mg oral dose
  Interventions: Drug: Alisporivir

INTERVENTIONS:
Drug: Alisporivir — Capsules supplied as open labeled bulk medication in 10-unit blister packages
  Other Names: DEB025

SUMMARY:
This is an open-label study to evaluate the pharmacokinetics, safety and tolerability of single oral doses of Alisporivir in subjects with mild and moderate hepatic impairment compared to matched healthy subjects with normal liver function.

ELIGIBILITY:
Inclusion criteria:

* Male or female, 18 to 70 years of age, in good health
* Stable Child-Turcotte-Pugh score of at least 5
* Body weight of at least 50 kg and a BMI of 18.0 to 36.0 kg/m2

Exclusion criteria:

* Use of other investigational drugs
* Women of child-bearing potential

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration (Cmax) of alisporivir | 0.5 h (± 5 min), 1 h (± 10 min), 2 h (± 10 min), 4 h (± 30 min), 6 h (± 30 min), 8 h (± 30 min), 12 h (± 30 min), 24 h (± 60 min), 48 h (± 60 min), 72 h (± 60 min), 96 h (± 60 min), 120 h (± 60 min), 144 h (± 60 min), and 168 h (± 60 min) post-dose
Area under the time-concentration curve (AUC) for alisporivir | 0.5 h (± 5 min), 1 h (± 10 min), 2 h (± 10 min), 4 h (± 30 min), 6 h (± 30 min), 8 h (± 30 min), 12 h (± 30 min), 24 h (± 60 min), 48 h (± 60 min), 72 h (± 60 min), 96 h (± 60 min), 120 h (± 60 min), 144 h (± 60 min), and 168 h (± 60 min) post-dose
  Categories: AUC up to the last measurable concentration (AUClast) and AUC from time 0 to the last time point measured (AUC0-t)

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) of alisporivir | 0.5 h (± 5 min), 1 h (± 10 min), 2 h (± 10 min), 4 h (± 30 min), 6 h (± 30 min), 8 h (± 30 min), 12 h (± 30 min), 24 h (± 60 min), 48 h (± 60 min), 72 h (± 60 min), 96 h (± 60 min), 120 h (± 60 min), 144 h (± 60 min), and 168 h (± 60 min) post-dose
Half-Life (T1/2) of alisporivir | 0.5 h (± 5 min), 1 h (± 10 min), 2 h (± 10 min), 4 h (± 30 min), 6 h (± 30 min), 8 h (± 30 min), 12 h (± 30 min), 24 h (± 60 min), 48 h (± 60 min), 72 h (± 60 min), 96 h (± 60 min), 120 h (± 60 min), 144 h (± 60 min), and 168 h (± 60 min) post-dose
Apparent total body clearance from plasma (CL/F) of alisporivir | 0.5 h (± 5 min), 1 h (± 10 min), 2 h (± 10 min), 4 h (± 30 min), 6 h (± 30 min), 8 h (± 30 min), 12 h (± 30 min), 24 h (± 60 min), 48 h (± 60 min), 72 h (± 60 min), 96 h (± 60 min), 120 h (± 60 min), 144 h (± 60 min), and 168 h (± 60 min) post-dose
Apparent volume of distribution (Vz/F) of alisporivir | 0.5 h (± 5 min), 1 h (± 10 min), 2 h (± 10 min), 4 h (± 30 min), 6 h (± 30 min), 8 h (± 30 min), 12 h (± 30 min), 24 h (± 60 min), 48 h (± 60 min), 72 h (± 60 min), 96 h (± 60 min), 120 h (± 60 min), 144 h (± 60 min), and 168 h (± 60 min) post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Novartis Institutes for BioMedical Research
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida